CLINICAL TRIAL: NCT06950775
Title: A Naturalistic Study of Residents of an Agriculturally Integrated Community
Brief Title: The Neighborhood & Health Study
Acronym: N&HS
Status: Recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY2025-0321
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy Eating; Cardiometabolic Health
Keywords: Agrihood; Physical Activity; Healthy Eating; Social Connectedness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Agrihood Group: The Agrihood Group consists of adults who live in the Indigo Neighborhood as their primary and permanent residence for less than 3 months or intend to move to the Indigo Neighborhood as their primary and permanent residence. Pregnant women will not be excluded from participation and may be coincidentally included.
  Interventions: Other: Residence in Agrihood Neighborhood
- Comparison Group: The Comparison Group consists of adults who live in the Elyson comparison neighborhood as their primary and permanent residence. Pregnant women will not be excluded from participation and may be coincidentally included.

INTERVENTIONS:
Other: Residence in Agrihood Neighborhood — We are examining the effects of individuals who move into an agrihood neighborhood.
  Groups: Agrihood Group

SUMMARY:
The objective of The Neighborhood & Health Study is to use a quasi-experimental mixed-methods approach to assess the impact of living in an agrihood-an agriculturally integrated community. This study follows a longitudinal cohort of residents of a newly developed neighborhood (the Indigo Neighborhood) and a geographically and socio-demographically matched neighborhood (the Elyson Neighborhood), both located in Fort Bend County, Texas, providing a unique opportunity for a natural experiment.

DETAILED DESCRIPTION:
Poor nutrition and inadequate physical activity are prevalent in many communities across the United States. Agriculturally integrated communities called "agrihoods" are a potential responsive agriculture solution that may support healthy living. The aims of the study are to 1) Assess short-term changes in healthy eating, physical activity, cardiometabolic health indicators, and social connectedness as compared to a comparison neighborhood that is not an agriculturally integrated neighborhood; 2) Document time use with features of the Indigo Agrihood and assess consumer preferences for built and nature design features to provide resident-driven data for future developments; 3) Assess the economic benefits of the Indigo Agrihood.

ELIGIBILITY:
Inclusion Criteria:

Indigo Neighborhood Participants:

* 18 years or older
* Lived in the Indigo Neighborhood as their primary and permanent residence for less than 3 months or intend to move to the Indigo Neighborhood as their primary and permanent residence.
* Pregnant women will not be excluded from participation and may be coincidentally included

Elyson Neighborhood Participants:

* 18 years or older
* Live in the Elyson Neighborhood as their primary and permanent residence (the comparison neighborhood group).
* Pregnant women will not be excluded from participation and may be coincidentally included

Exclusion Criteria:

Indigo Neighborhood Participants:

• None.

Elyson Neighborhood Participants:

• None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population the groups will be selected from are residents of the Indigo Neighborhood and Elyson Neighborhood in Fort Bent County, Texas
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in healthy eating | Baseline to 3 & 6 months
  Healthy eating will be measured by the Mediterranean Eating Pattern for Americans - 16 items scale. Score ranges from 0 to 16. Higher scores indicate healthy eating patterns.
Change in physical activity | Baseline to 3 & 6 months
  Physical activity will be measured through calculating moderate to vigorous physical activity (MVPA), light, moderate, and vigorous physical activity (LMVPA), walking, and sedentary behavior using data from an accelerometer worn by participants for 7 days
Change in body mass index (BMI) | Baseline to 6 months
  Height and weight will be measured by research staff and BMI will be calculated.
Change in blood pressure | Baseline to 6 months
  Blood pressure will be measured by research staff using an Omron sphygmomanometer. Measured in units of millimeters of mercury (mmHg).
Change in hemoglobin A1c | Baseline to 6 months
  Hemoglobin A1c will be measured by research staff using a CardioChek Plus machine that measures glucose in their blood. Hemoglobin A1c is measured in milligrams (mg) per deciliter (dL) of blood.
Change in social connectedness | Baseline to 3 & 6 months
  Social connectedness will be measured by the Brief Sense of Community Scale. Scores range from 8 to 40. Higher scores indicate more social connectedness.

SECONDARY OUTCOMES:
Change in total physical activity | Baseline to 3 & 6 months
  Total physical activity (MET-min/wk) will be assessed using the International Physical Activity Questionnaire short form (IPAQ-long)
Change in dermal carotenoids | Baseline to 6 months
  Dermal carotenoids will be measured by research staff using a Veggie Meter machine, which scans a participant's finger to measure carotenoids or how many fruits and vegetables someone eats. Scores from 0 to 800. Higher scores indicate higher levels of carotenoids.
Change in lipids | Baseline to 6 months
  Lipids will be measured by research staff using a CardioChek Plus machine that measures lipids in blood. Triglycerides will be measured in milligrams (mg) of triglycerides per deciliter (dL) of blood. LDL/HDL cholesterol will be measured in milligrams of LDL/HDL cholesterol per deciliter (dL) of blood. Total Cholesterol is measured in milligrams (mg) of cholesterol per deciliter (dL) of blood.
Change in total HEI score | Baseline to 3 & 6 months
  Total Healthy Eating Index (HEI) score will be calculated from a single 24-hour recall collected via the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). Score ranges from 0 to 100. Higher scores indicate better diet.
Change in fruit intake | Baseline to 3 & 6 months
  Total fruit intake (cups/day) will be measured using a LS7 item.
Change in vegetable intake | Baseline to 3 & 6 months
  Total vegetable intake (cups/day) will be measured using a LS7 item.
Change in consumption of whole grains | Baseline to 3 & 6 months
  Whole grain consumption (servings/day) will be assessed using an LS7 item.
Change in fiber intake | Baseline to 3 & 6 months
  Fiber intake (g/day) will be assessed using the NHANES Dietary Screener Questionnaire (DSQ).
Met recommendation for fish consumption (y/n) | Baseline to 3 & 6 months
  Whether or not a participant met the recommendation for fish consumption will be assessed using an LS7 item.
Change in frequency of consuming ultra-processed foods | Baseline to 3 & 6 months
  Frequency of ultra-processed foods consumption (times/month) will be assessed using a 9-item questionnaire adapted from the DSQ and the Beverage and Snack Questionnaire (BSQ2).
Change in red and processed meat consumption | Baseline to 3 & 6 months
  Total red and processed meat consumption (g/week) will be estimated using the DSQ.
Change in alcohol consumption | Baseline to 3 & 6 months
  Alcohol consumption (drinks/day) will be assessed using a 2-item questionnaire adapted from the Alcohol Use Disorders Screening Test (AUDIT).
Change in American Heart Association's Life's Simple 7 (LS7) cardiovascular health score | Baseline to 3 & 6 months
  American Heart Association's Life's Simple 7 (LS7) score is a composite of cardiovascular disease (CVD) risk factors (physical activity, eating habits, smoking status, cholesterol, glucose, body mass index (BMI), and blood pressure). Score ranges from 0 to 14. Higher scores indicate better health.
Change in World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) recommendation adherence score | Baseline to 3 & 6 months
  WCRF/AICR recommendation adherence score is a composite of seven items listed above: BMI, physical activity, fiber intake, fruit and vegetable consumption, processed food consumption, red meat consumption, and alcohol consumption. Scores range from 0 to 7. Higher scores indicate greater adherence to the recommendations.
Change in American Heart Association's Life's Essential 8 (LE8) cardiovascular health score | Baseline to 3 & 6 months
  American Heart Association's Life's Essential 8 (LE8) score is a composite of cardiovascular disease (CVD) risk factors (physical activity, eating habits, smoking status, sleep, cholesterol, glucose, body mass index (BMI), and blood pressure). Score ranges from 0 to 100. Higher scores indicate better health.
Change in community food environment | Baseline to 3 & 6 months
  The community food environment, including store access and shopping behaviors, will be assessed by two items from the Perceived Nutrition Environment Measures Survey. Scores range from 2 to 10. Higher scores indicate a more diverse community food environment
Change in perceived stress | Baseline to 3 & 6 months
  Perceived stress will be assessed by the Perceived Stress Scale. Scores range from 0 to 40. Higher scores indicate more perceived stress.
Change in gardening and fruit and vegetable procurement | Baseline to 3 & 6 months
  Types of gardening and where fruits and vegetables are obtained will be assessed using multiple choice questions.
Change in sense of community | Baseline to 3 & 6 months
  Sense of community will be assessed using the Collective Efficacy scale. Scores range from 5 to 25. Higher scores indicate greater sense of community.
Change in nature exposure | Baseline to 3 & 6 months
  Nature exposure will be assessed by modified questions from the People and Nature Survey for England for American audiences. Multiple choice questions assess how much time is spent in nature and what type of natural spaces individuals visit. An additional multiple-choice item from the Nature of Americans survey will be used to identify how much time is spent in nature recreationally and for work in a typical week in hours.
Change in positive and negative affect | Baseline to 3 & 6 months
  Positive and negative affect will be assessed by the Positive and Negative Affect Scale. Scores range from 10 to 50 for each positive and negative affect. Higher scores indicate more positive or negative affect.
Change in (community) social cohesion | Baseline to 3 & 6 months
  Community social cohesion will be assessed by the social cohesion sub-scale of the Mujahid et al. Neighborhood Environment Scale (NES). Scores range from 1 to 5. Higher scores indicate greater social cohesion.
Change in transportation used to utilized food resources | Baseline to 3 & 6 months
  Transportation used to obtain food will be assessed by a single categorical item.
Change in distance to utilized food resources | Baseline to 3 & 6 months
  Distance to utilized food resources will be measured in miles.
Change in number of utilized food resources | Baseline to 3 & 6 months
  Number of utilized food resources will be measured by a multiple choice item.
Change in transportation used to utilized physical activity resources | Baseline to 3 & 6 months
  Transportation used to access the physical activity resources will be assessed by a single categorical item.
Change in distance to utilized physical activity resources | Baseline to 3 & 6 months
  Distance to utilized physical activity resources will be measured in miles.
Change in number of utilized physical activity resources | Baseline to 3 & 6 months
  Number of utilized physical activity resources will be measured by a multiple choice item.
Change in loneliness | Baseline to 3 & 6 months
  Loneliness and social isolation will be assessed by the UCLA Loneliness Scale. Scores range from 20 to 80. Higher scores indicate more loneliness and social isolation.
Change in functional health | Baseline to 3 & 6 months
  Functional health will be assessed by the Quality Metric's MOS Short Form - 36 Version 2. 10 items will be used with scores range from 0 to 20. Higher scores indicate higher functional health.
Change in fruit intake | Baseline to 3 & 6 months
  Total fruit intake (cups/day) will be measured using a 24-hour recall.
Change in vegetable intake | Baseline to 3 & 6 months
  Total vegetable intake (cups/day) will be measured using a 24-hour recall.
Change in consumption of whole grains | Baseline to 3 & 6 months
  Whole grain consumption (servings/day) will be assessed using a 24-hour recall.
Change in fiber intake | Baseline to 3 & 6 months
  Fiber intake (g/day) will be assessed using a 24-hour recall.
Change in red and processed meat consumption | Baseline to 3 & 6 months
  Total red and processed meat consumption (g/week) will be estimated using a 24-hour recall.
Change in alcohol consumption | Baseline to 3 & 6 months
  Alcohol consumption (drinks/day) will be assessed using a 24-hour recall.
Change in frequency of consuming ultra-processed foods | Baseline to 3 & 6 months
  Frequency of ultra-processed foods consumption (times/month) will be assessed using a 24-hour recall.

CONTACTS AND LOCATIONS:
Overall Officials: Jay E Maddock, Ph.D., Principal Investigator — Texas A&M University
Locations (2):
- United States (2):
  - Elyson Neighborhood, Katy, Texas
  - Indigo Neighborhood, Richmond, Texas

REFERENCES:
- [Derived] Maddock JE, Lewis EC, Villarreal DL, MacMillan Uribe AL, Janda-Thomte KM, Han G, Hall CR, Sturdivant RX, Patterson MS, Graham ML, Seguin-Fowler RA, Umstattd Meyer MR. Protocol for a naturalistic study of residents living in an agriculturally-integrated ("agrihood") neighborhood. Front Public Health. 2025 Nov 20;13:1679602. doi: 10.3389/fpubh.2025.1679602. eCollection 2025. PMID 41358215